CLINICAL TRIAL: NCT05481671
Title: Influencing Factors and Their Approach of Kinesiophobia in Patients With Traumatic Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: kinesiophobia（fracture)2022.07
Record Dates: First submitted 2022-07-24; First posted 2022-08-01 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Traumatic Fracture
Keywords: Traumatic Fracture; Kinesiophobia; Pain Catastrophizing; Anxiety; Depression; Self-efficacy; Psychological Resilience
MeSH Terms: conditions — Kinesiophobia; Anxiety Disorders; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Study subjects are hospitalized patients with traumatic fractures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires assessed patients with traumatic fractures: ①Age 18 and above.
  ②Patients who were diagnosed as fractures due to accidental trauma and were diagnosed by X-rays and clinicians and required surgical treatment.
  ③Have the normal cognitive ability, expression ability and social participation ability.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Participants will be asked to respond to the Demographic Information Sheet, Tampa Scale for Kinesiophobia, Numeric Rating Scale, Pain Catastrophizing Scale, Hospital Anxiety and Depression Scale, Resilience Scale , Pain Self-efficacy Questionnaires and Functional Exercise Compliance Scale for Orthopaedic Patients.

SUMMARY:
This study aims to investigate the relationship between kinesiophobia and pain catastrophizing, as well as the relationship between pain catastrophizing and pain level, anxiety and depression, self-efficacy and psychological resilience in patients with traumatic fractures, and to explain the approach and effect relationship between kinesiophobia and these variables.

DETAILED DESCRIPTION:
At present, there are few studies on kinesiophobia in patients with traumatic fractures. This study adopts structural equation model to analyze the current situation of kinesiophobia in patients with traumatic fractures, and explores the effect of pain level, pain catastrophizing, anxiety and depression, self-efficacy and psychological resilience on kinesiophobia in patients with traumatic fractures, which provides a scientific basis for predicting the occurrence of kinesiophobia in patients with traumatic fractures and developing intervention plans.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as fractures due to accidental trauma and were diagnosed by X-rays and clinicians and required surgical treatment.
* Age 18 and above.

Exclusion Criteria:

* Those with a history of chronic pain (pain persisting or indirectly persisting for more than 3 months).
* Those who have serious postoperative complications (such as deep vein thrombosis, infection, etc.) and need other treatment or transfer to another department.
* People with physical disability or abnormal muscle strength before injury.
* Those who have a history of mental illness or who have taken anti-anxiety, depression drugs, or cognitive impairment within one month.
* Patients undergoing emergency surgery on the day of admission.
* Those who cannot communicate normally due to physical or psychological barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients with traumatic fractures admitted to the Orthopedics Department of the three third-class hospitals in Guangzhou from August 2022 to May 2023.
Sampling Method: Non-Probability Sample
Enrollment: 381 (Estimated)
Dates: Start 2022-10-02 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
kinesiophobia | baseline
  The kinesiophobia level of patients with traumatic fractures will be measured by Tampa Scale for Kinesiophobia（TSK-11）. The total score ranges from 11 to 44. A score of more than 26 on the scale is defined as kinesiophobia.
kinesiophobia | 3 days after surgery
  The kinesiophobia level of patients with traumatic fractures will be measured by Tampa Scale for Kinesiophobia（TSK-11）. The total score ranges from 11 to 44. A score of more than 26 on the scale is defined as kinesiophobia.
functional exercise compliance | 3 days after surgery
  The compliance of functional exercise in patients with traumatic fractures will be measured by Functional Exercise Adherence Scale for Orthopaedic Patients. The total score ranges from 15 to 75. A total score of less than or equal to 20 indicates low compliance; a score of greater than or equal to 55 indicates high compliance; and a score of greater than 20 and less than 50 indicates partial compliance.

SECONDARY OUTCOMES:
pain degree | baseline
  The pain degree of patients with traumatic fractures will be measured by Numberical Rating Scale. Pain is scored on a scale of 0 to 10, with higher scores indicating higher pain degree.
pain degree | 3 days after surgery
  The pain degree of patients with traumatic fractures will be measured by Numberical Rating Scale. Pain is scored on a scale of 0 to 10, with higher scores indicating higher pain degree.
pain catastrophization | baseline
  The level of catastrophic pain in patients with traumatic fractures will be measured by Pain Catastrophizing Scale. Scores range from 0 to 52, with higher scores indicating higher levels of catastrophic pain in patients.
pain catastrophization | 3 days after surgery
  The level of catastrophic pain in patients with traumatic fractures will be measured by Pain Catastrophizing Scale. Scores range from 0 to 52, with higher scores indicating higher levels of catastrophic pain in patients.
anxiety and depression | baseline
  The anxiety and depression of patients with traumatic fractures will be measured by Hospital Anxiety and Depression Scale . The scale score ranges from 0 to 21 points, 0 to 7 points for no anxiety or depression, 8 to 10 points for suspicious symptoms of anxiety or depression, and greater than or equal to 11 points for psychological disorders.
anxiety and depression | 3 days after surgery
  The anxiety and depression of patients with traumatic fractures will be measured by Hospital Anxiety and Depression Scale . The scale score ranges from 0 to 21 points, 0 to 7 points for no anxiety or depression, 8 to 10 points for suspicious symptoms of anxiety or depression, and greater than or equal to 11 points for psychological disorders.
self-efficacy | baseline
  The self-efficacy of patients with traumatic fractures will be measured by Pain Self-efficacy Scale. The total score ranges from 0 to 60, with higher scores indicating higher pain self-efficacy.
self-efficacy | 3 days after surgery
  The self-efficacy of patients with traumatic fractures will be measured by Pain Self-efficacy Scale. The total score ranges from 0 to 60, with higher scores indicating higher pain self-efficacy.
psychological resilience | baseline
  The psychological resilience of patients with traumatic fractures will be measured by Resilience Scale (CD-RISC-10). The total score ranges from 0 to 40, with higher scores indicating higher psychological resilience.
psychological resilience | 3 days after surgery
  The psychological resilience of patients with traumatic fractures will be measured by Resilience Scale (CD-RISC-10). The total score ranges from 0 to 40, with higher scores indicating higher psychological resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No